CLINICAL TRIAL: NCT04241952
Title: Effects of Early Exercise in Patients With Moderate to Severe Stroke - a Randomized Controlled Trial
Brief Title: Effects of Early Exercise in Patients With Moderate to Severe Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klas Sandberg (Other)
Responsible Party: Sponsor-Investigator, Klas Sandberg, Clinical Investigator, Ostergotland County Council, Sweden
Organization: Ostergotland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stroke2015
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Exercise; Bedcycling
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Usual care and bedcycling.
  Interventions: Other: Exercise
- Control group (No Intervention): Usual care

INTERVENTIONS:
Other: Exercise — Bedcycling
  Arms: Exercise group

SUMMARY:
Purpose: to investigate the efficacy of early exercise in patients with moderate to severe stroke regarding functional outcome and walking ability.

Methods: Patients with medium to severe stroke (NHISS >7) were recruited 24 - 48 hours after stroke onset from two stroke units in Sweden. Both groups received usual care. The intervention group received even 20 minutes bed-cycling 5 days per week with a maximum of 15 sessions. Functional outcome was measured with modified Rankin Scale (mRS) and Barthel index and walking with the 6-minute walking test (6MWT). Measurements were performed pre- and post-intervention (3 weeks), and at 3-months follow-up.

ELIGIBILITY:
Inclusion criteria:

* Age over 18 years.
* Diagnose stroke with The National Institutes of Health Stroke Scale (NIHSS) 7-42 points.
* Ability to understand the Swedish language.
* Approval of medical responsible physician to participate in the study.

Exclusion criteria:

• Medical or neurological diseases that can affect the performance of the exercise and severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Modified Rankin Scale (mRS) | Baseline 24-48 hours after onset, postintervention 3 weeks after baseline and follow up 3-months after baseline.
  Functional Outcome

SECONDARY OUTCOMES:
Change in Barthel ADL-Index | Baseline 24-48 hours after stroke onset, postintervention 3-weeks after baseline and follow up 3-months after baseline.
  ADL
Change in 6-Minutes Walking test (6MWT) | Baseline 24-48 hours after stroke onset, postintervention 3-weeks after baseline and follow up 3-months after baseline.
  Walking Ability

CONTACTS AND LOCATIONS:
Overall Officials: Paul Enthoven, PhD, Principal Investigator — Linkopings University,Sweden

REFERENCES:
- [Derived] Sandberg K, Kleist M, Enthoven P, Wijkman M. Hemodynamic responses to In-Bed Cycle Exercise in the acute phase after moderate to severe stroke: A randomized controlled trial. J Clin Hypertens (Greenwich). 2021 May;23(5):1077-1084. doi: 10.1111/jch.14232. Epub 2021 Mar 11. PMID 33704913